CLINICAL TRIAL: NCT07288918
Title: The Effects of Different Educational Methods Given to Patients Undergoing Organ Transplantation on Quality of Life, Compliance With İmmunosuppressive Therapy and Symptom Control
Brief Title: The Effect of Education on Quality of Life, Adherence to Immunosuppressive Therapy and Symptom Control in Organ Transplant Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Rıfat GÜRKAN, Principal Investigator, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OMU-GURKAN-001
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Organ Transplantation; Mobile Applications; Nursing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mobile applications (Experimental)
  Interventions: Other: Mobile application installation
- Teaching booklet (Experimental)
  Interventions: Other: Providing teaching booklets
- Control (Active Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Other: Mobile application installation — Transplant patients will receive standard discharge training. A mobile application created by the researcher will be installed on transplant patients' phones.
  Arms: Mobile applications
Other: Providing teaching booklets — Transplant patients will receive standard discharge training. Transplant patients will be given researcher prepared instructional booklet
  Arms: Teaching booklet
Other: Control — Transplant patients will receive standard discharge training
  Arms: Control

SUMMARY:
Organ transplantation is the most effective method for treating end-stage organ failure and allows patients on the verge of death to continue living. Organ transplantation involves removing all or part of an organ or tissue from the body and transplanting it to suitable patients experiencing failure. Therefore, transplants are performed to treat diseases, save lives, improve patients' quality of life, and extend their life expectancy. The World Health Organization (WHO) defines quality of life as individuals' perceptions of their goals, expectations, standards, and concerns regarding their place in life, within the context of the culture and value systems they live in. Achieving an adequate quality of life after transplantation is considered an indicator of therapeutic success, which is increasingly important to measure by the transplant care team.

Individuals who undergo transplantation and their families often perceive transplantation as a rebirth. However, 30% to 40% of patients report no better health-related quality of life after kidney transplantation compared to dialysis. This is attributed to frequent checkups and monitoring, new medications and their strict dosing schedules, and the unexpected discomfort of potential side effects.

Even after the psychological challenges of waiting and the joy of a successful transplant, transplant recipients take on new responsibilities. Problems such as accepting transplantation risks, acute and chronic organ rejection, and adherence to lifelong medication regimens can arise. Persistent side effects of various immunosuppressive agents, adaptation and maintenance of the new organ, and uncertainty about the future due to rejection of transplanted organs and the subsequent re-transplantation process can all lead to physical and psychological distress.

Immunosuppressive therapy represents a lifelong endeavor for transplant recipients. These medication regimens involve complex protocols, not only due to the number of pills required, but also due to blood level monitoring, side effects, and frequent dose adjustments to avoid rejection. Non-adherence to immunosuppressant regimens has been shown to be high in organ transplant patients. Non-adherence rates in this population are reported as high as 65%. The highest immunosuppressant non-adherence rate is found in kidney transplant recipients, with a prevalence of 36-55%, while this rate is 15-40% in liver transplant recipients. Studies have found that 16-36% of graft losses are associated with non-adherence. The ever-growing population of transplant recipients and the limited number of transplant centers, particularly those living farther away, necessitate innovative healthcare delivery models to monitor and improve the use of transplant center resources. With the advent of smartphones and mobile medical devices, mobile health has become a popular way for healthcare professionals to manage patient care. Mobile health can serve as an adjunct method for delivering health education information, sending reminders to patients to take their medications, and implementing online education. In particular, converting paper-based education to video format can significantly increase knowledge on various topics. It is necessary to address the problems and challenges patients face after discharge and the practices that can potentially address these issues. These results suggest that healthcare professionals can do more to provide comprehensive care to patients, promote successful home-based treatment regimens, symptom control, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age,
* Having undergone a liver or kidney transplant for the first time,
* Having been discharged at least three months ago,
* Having access to a smartphone and internet and the ability to use them independently,

Exclusion Criteria:

* Having a diagnosis of a psychiatric or neurological disorder,
* Having hearing or vision problems severe enough to impede communication,
* Requesting to leave during the research period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
The effect of education on quality of life in organ transplant patients | Baseline, and 1, 3, and 6 months post-intervention.
  The SF-36 Quality of Life Scale will be administered before the training intervention. Most questions on the scale use Likert-type rating scales (3, 5, and 6 points), while questions four and five can be answered with yes/no. Each section of the scale is rated between 0 and 100 points. Higher scores indicate better health, or improved quality of life ("0" for poor health, "100" for good health).
The effect of education on symptom control in organ transplant patients | Baseline, and 1, 3, and 6 months post-intervention.
  The Modified Transplant Symptom Occurrence and Symptom Distress Scale-59 will be administered before the training intervention. Each item on the scale corresponds to a side effect of immunosuppressive drugs, and these items have two dimensions that assess symptom occurrence and discomfort level. Symptom occurrence is scored from 1 to 5, with 1=never occurring and 5=always occurring. Symptom discomfort level is scored from 0 to 4, with 0=never causing discomfort and 4=causing extreme discomfort.
The effect of education on adherence to ımmunosuppressive therapy in organ transplant patients | Baseline, and 1, 3, and 6 months post-intervention.
  The Immunosuppressant Therapy Adherence Scale in Organ Transplantation Patients will be administered before the training intervention. The scale consists of four questions, and participants can receive a score between 0 and 12. Individuals who have not forgotten their immunosuppressive treatment in the last three months are given 3 points, those with 1-20% non-adherence to immunosuppressive treatment are given 2 points, those with 21-50% non-adherence to immunosuppressive treatment are given 1 point, and those with >50% non-adherence to immunosuppressive treatment are given 0 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayis University, Samsun, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No